CLINICAL TRIAL: NCT02149342
Title: Daylight-mediated Photodynamic Therapy of Actinic Keratoses: a Randomized, Double-blinded Pilot Study Comparing Topical 0.2% Hexylaminolaevulinate With 16% Methylaminolaevulinate
Brief Title: Daylight-mediated Photodynamic Therapy of Actinic Keratoses:Comparing 0.2%HAL With 16%MAL
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Joint Authority for Päijät-Häme Social and Health Care (Other)
Collaborators: Helsinki University Central Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 2013-001389-40
Record Dates: First submitted 2014-05-19; First posted 2014-05-29 (Estimated); Results first posted 2016-07-11 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-05

CONDITIONS: Actinic Keratoses
Keywords: Actinic keratoses; Daylight-PDT; Hexylaminolaevulinate; HAL; Methylaminolaevulinate; MAL; Hyperspectral imaging
MeSH Terms: conditions — Keratosis, Actinic | interventions — 5-aminolevulinic acid hexyl ester; methyl 5-aminolevulinate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- HAL cream and MAL cream (Experimental): 0.2% HAL (Hexvix, Photocure) mixed with Unguentum M (Allmiral) and MAL (Metvix, Galderma) used in a randomized split-face design
  Interventions: Drug: Hexylaminolaevulinate cream; Drug: Methylaminolaevulinate cream

INTERVENTIONS:
Drug: Hexylaminolaevulinate cream — 0.2% Hexylaminolaevulinate (Hexvix, Photocure) mixed with Unguentum M (Allmiral) cream (2014)
  Other Names: HAL; Hexvix, Photocure
Drug: Methylaminolaevulinate cream — MAL 16% is used as photosensitizer for daylight-PDT
  Other Names: 16% Methylaminolaevulinate (Metvix, Galderma) cream; MAL

SUMMARY:
This pilot study compares two photosensitizers, hexylaminolaevulinate (HAL) and methylaminolaevulinate (MAL), in treatment of actinic keratoses. Study is conducted using randomized split-face design. Efficacy is assessed clinically, and histologically at 3 and 12 months. Pain during and after treatments and adverse reactions at one week are recorded.

DETAILED DESCRIPTION:
Study recruites 16-20 voluuntering patients with symmetrical actinic damage on face or scalp. Treatment sites are randomized to receive either hexylaminolaevulinate 0.2% or methylaminolaevulinate ( 16% MAL) as photosensitizers (0.25mm-thick layer). A web-based validated program (Research Randomizer) generated a randomized list to define the treatment sides. The randomization results were kept blinded from the investigators who conducted the follow-up visits, from the pathologist, and the patients. Pre-treatment procedures include application of sunscreen for 15 minutes and curettage of the treatment area. Illumination is performed using 2 hours daylight-exposure. Efficacy is assessed clinically, and histologically at 3 and 12 months by blinded observers. Pain during and after treatments and adverse reactions at one week are recorded.

ELIGIBILITY:
Inclusion Criteria:

-Symmetrical actinic damage on face or scalp

Exclusion Criteria:

* Pregnancy
* Lactation
* Allergy to photosensitizer
* Photodermatose

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2014-05; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Noora E Neittaanmäki-Perttu, MD, Principal Investigator — Päijät-Häme Cnetral Hospital, Helsinki University Central Hospital; Mari Grönroos, MD, PhD, Study Director — Päijät Häme Central Hospital
Locations (1):
- Päijät-Häme Central Hospital, Lahti, Lahti, Finland

IPD SHARING:
Plan to Share IPD: Yes
International peer-reviewed publication

REFERENCES:
- [Result] Neittaanmaki-Perttu N, Gronroos M, Karppinen TT, Tani TT, Snellman E. Hexyl-5-aminolaevulinate 0.2% vs. methyl-5-aminolaevulinate 16% daylight photodynamic therapy for treatment of actinic keratoses: results of a randomized double-blinded pilot trial. Br J Dermatol. 2016 Feb;174(2):427-9. doi: 10.1111/bjd.13924. Epub 2015 Nov 20. No abstract available. PMID 26011755

RESULTS

PARTICIPANT FLOW:
Groups:
- Hexylaminolaevulinate and Methylaminoalevulinate Creams: 0,2% hexylaminolaevulinate cream , HAL (Hexvix, Photocure, Unguentum M, Almirall) 16% methylaminolaevulinate, MAL (Metvix, Galderma)
  HAL and MAL used as photosensitizer for daylight-PDT in a randomized split-face design
Period: Overall Study
Arm/Group | Hexylaminolaevulinate and Methylaminoalevulinate Creams
Started | 14 (14 patients)
Completed | 14 (14 patients)
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Hexylaminolaevulinate and Methylaminoalevulinate Cream: 0.2% hexylaminolaevulinate (Hexvix, Photocure) mixed with Unguentum M (Allmiral) and 16% methylaminolaevulinate (Metvix, Galderma) in a split-face design
Arm/Group | Hexylaminolaevulinate and Methylaminoalevulinate Cream
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 14
Age, Continuous [Mean (Full Range); unit: years] | 79 [66 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 6
Region of Enrollment [Number; unit: participants]
  Finland | 14

OUTCOME MEASURES:

1. Primary Outcome: Histological Lesion Clearance
Description: Punch biopsies were taken symmetrically on both treatment fields from equally graded >6 mm AKs prior to treatment and again at 3 months, blinded observer (pathologist). HE- and p53-stainings. Samples not fulfilling the criteria of an AK were defined as healthy or completely cleared. The p53 reactivity expressed as average percentage of positive nuclei in three consecutive high power fields from the region of highest reactivity (<10 % normal)
Time Frame: Baseline, 3 months
Population: One patient was excluded from the histological analysis because one biopsied lesion clinically taken as an AK appeared histologically to be seborrheic eczema.
Measure: Mean (Full Range); unit: percentage of complete histological clea
Units Other Than Participants: Punch biopsies
Groups:
- Hexylaminolaevulinate Cream: 0.2% hexylaminolaevulinate (Hexvix, Photocure) mixed with Unguentum M (Allmiral)
  Hexylaminolaevulinate cream: 0.2% Hexylaminolaevulinate (Hexvix, Photocure) mixed with Unguentum M (Allmiral) cream
- Methylaminolaevulinate Cream: 16% methylaminolaevulinate (Metvix, Galderma)
  Methylaminolaevulinate cream: MAL 16% is used as photosensitizer for daylight-PDT
Arm/Group | Hexylaminolaevulinate Cream | Methylaminolaevulinate Cream
Number analyzed (Participants) | 13 | 13
Number analyzed (Punch biopsies) | 26 | 26
percentage of complete histological clea | 38.5 [0 to 100] | 69.2 [0 to 100]

2. Secondary Outcome: Clinical Lesion Clearance
Description: Clinical lesion clearance is observed by a blinded observer
Time Frame: Baseline, 3 months
Measure: Mean (Full Range); unit: percentage of lesions in complete respon
Units Other Than Participants: AK lesions
Groups:
- Hexylaminolaevulinate Cream: 0.2% hexylaminolaevulinate (Hexvix, Photocure) mixed with Unguentum M (Allmiral) (2014) 2% hexylaminolaevulinate (Hexvix Photocure) mixed with Unguentum M (Allmiral) (2015)
  Hexylaminolaevulinate cream: 0.2% Hexylaminolaevulinate (Hexvix, Photocure) mixed with Unguentum M (Allmiral) cream (2014)
Arm/Group | Hexylaminolaevulinate Cream | Methylaminolaevulinate Cream
Number analyzed (Participants) | 14 | 14
Number analyzed (AK lesions) | 103 | 98
percentage of lesions in complete respon | 73.4 [28.6 to 100] | 77.8 [44.4 to 100]

3. Secondary Outcome: Adverse Reactions
Description: Adverse reactions are evaluated by blinded observer at one week after treatment. Severity of the reaction ( Redness, crusting and scaling) is assessed using grading: minimal, mild, intermediate, severe.
Time Frame: One week
Measure: Number; unit: participants
Arm/Group | Hexylaminolaevulinate Cream | Methylaminolaevulinate Cream
Number analyzed (Participants) | 14 | 14
participants | 14 | 14

4. Secondary Outcome: Pain Assesment (Visual Analog Scale)
Description: Pain using visual analog scale (VAS 0-10, where 0 is no pain and 10 is the worst pain imaginable) on both treatment sides is assessed in every 30 minutes during 2-hour sun-exposure and afterwards once in two hours until 9 p.m. (treatment day). Of these values, the mean maximal pain is assessed.
Time Frame: 12 hours
Measure: Mean (Full Range); unit: Mean maximal pain VAS score
Arm/Group | Hexylaminolaevulinate Cream | Methylaminolaevulinate Cream
Number analyzed (Participants) | 14 | 14
Mean maximal pain VAS score | 0.86 [0.1 to 2.2] | 1 [0.1 to 4.4]

5. Other Pre Specified Outcome: Clearance of Field Cancerization in Hyperspectral Images
Description: Data not collected
Time Frame: 3 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse reactions were assessed by blinded observer at one week after treatment Cosmetic outcome was evaluated at 3 months
Arm/Group | Hexylaminolaevulinate Cream | Methylaminolaevulinate Cream
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 14/14 | 14/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hexylaminolaevulinate Cream (N=14) | Methylaminolaevulinate Cream (N=14)
Redness, crusting, scaling; minimal (Skin and subcutaneous tissue disorders) | 10 (10) | 3 (3)
Redness, scaling, crusting; Mild (Skin and subcutaneous tissue disorders) | 3 (3) | 9 (9)
Redness, crusting, scaling; intermediate (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Redness, scaling, crusting; Severe (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
As the study was conducted as a single center pilot study, the results should be confirmed in a larger trial also valuing the patient complete response rates. A further limitation was we did not record light-doses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No